CLINICAL TRIAL: NCT03137264
Title: An Open-Label, Non-randomized, Prospective Biomarker Study to Assess Analytic Concordance Between Non-invasive Testing and Tissue Testing for EGFR T790M Mutation Detection in Patients With Non-small Cell Lung Cancer
Brief Title: Resistance & Activating Mutations Diagnosed Among NSCLC Community Dwelling EGFR Mutation Positive Patients
Acronym: RADIANCE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: D5160L00032
Record Dates: First submitted 2017-04-20; First posted 2017-05-02 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: T790M mutation; EGFR epidermal growth factor receptor; non-invasive testing; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, urine, and tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- T790M positive: Patients determined to be T790M positive on cobas tissue and/or cobas plasma testing during Part 1 may be followed for clinical outcomes in Part 2, and will be treated in accordance with standard of care, which may include osimertinib.
  Interventions: Drug: Other
- T790M negative: Patients determined to be T790M negative during Part 1 will not be followed for clinical outcomes in Part 2.

INTERVENTIONS:
Drug: Other — Patients who are T790M positive via cobas plasma and/or cobas tissue testing during Part 1 will be treated per standard of care during Part 2, which may include osimertinib.
  Other Names: Standard of Care
  Groups: T790M positive

SUMMARY:
The study is being done to determine if non-invasive testing (urine and plasma testing) is as effective as tissue testing in identifying epidermal growth factor receptor (EGFR) T790M mutation status. EGFR is a type of protein found on the surface of cells in the body. When this protein is mutated and becomes too active, it can lead to cancer growth. T790M is a mutation that develops in response to treatment of the EGFR mutation.

Participating patients will have tumor tissue (via cobas test), as well as 2 plasma samples (via cobas and Guardant360 tests) and 1 urine sample (via Trovera test), tested for EGFR T790M mutation status. If the results of the cobas tissue and/or plasma test show that a patient is T790M positive, they will be treated according to standard of care, which may include treatment with osimertinib. Osimertinib is approved for use in the United States for the treatment of EGFR T790M mutation-positive non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
RADIANCE is an open-label, prospective biomarker study to assess analytic concordance between non-invasive testing (plasma and urine) and tissue testing for the EGFR T790M mutation. All patients will have tumor tissue (via cobas test) as well as 2 plasma samples (via cobas and Guardant360) and 1 urine sample (via Trovera) tested for the EGFR T790M mutation (Part 1). Patients who are confirmed T790M negative based on both cobas biomarker tests (tissue and plasma) will have completed the study. Patients who demonstrate T790M+ on cobas tissue and/or cobas plasma testing may choose to undergo treatment with osimertinib in consultation with their healthcare provider (no investigational product will be provided for this study) and will continue to Part 2. In case of insufficient samples for biomarker testing or invalid results from any of the 4 testing modalities, another sample may be acquired from the patient, if feasible, including the patient's decision to undergo a second biopsy. Failure of a patient to undergo a tissue, plasma, or urine sample collection for biomarker testing will result in their withdrawal from the study. If 1 or more samples are insufficient for testing or 1 or more of the test results are invalid, the patient may still qualify for the clinical outcomes part of the study (Part 2) as long as cobas tissue and/or cobas plasma test is T790M+ and the patient receives at least one dose of osimertinib.

During Part 2 Follow-Up Visits will occur according to standard of care, but at least every 12 weeks for the first 12 months of treatment. A Final Study Visit will occur at 18 months (Week 72 +/- 14 days) or upon early withdrawal.

Statistical methods Sample size: The sample size is such to provide enough statistical precision for the primary endpoint. A sample size of 400 patients with evaluable biomarker test results for analytic concordance has been selected in order to achieve a precision of no more than ±5% around the estimated concordance rate. If a 15% inflation factor is applied (~70 patients) to this sample size to take into account those patients who may not be evaluable for concordance estimates, a total of approximately 470 patients will be enrolled.

The Full Analysis Sets will include the following:

Part 1: All patients in the study with cobas tissue, Guardant360 plasma, and Trovera urine test results.

Part 2: Patients who demonstrate T790M+ cobas tissue and/or cobas plasma testing and were treated with at least 1 dose of osimertinib (i.e., all patients in Part 2).

Safety analysis sets: The safety analysis sets will include the following:

Part 1: All patients in the study from the time of informed consent until completion of Part 1.

Part 2: Patients who demonstrate T790M+ cobas tissue and/or cobas plasms testing and were treated with at least 1 dose of osimertinib (i.e., all patients in Part 2).

The analyses of the data collected within this study will be descriptive only, with no formal statistical testing. Continuous variables will be summarized by the number of observations, mean, standard deviation, median, minimum, and maximum. Categorical variables will be summarized by frequency counts and percentages for each category. A Statistical Analysis Plan will be prepared and finalized prior to the first interim analysis, which will occur upon completion of the diagnostic analytic validity part of the study (Part 1). The concordance rate between non-invasive testing and cobas tissue testing will be presented as the point estimate together with the exact 95% confidence interval (CI) estimated using the Clopper-Pearson method. The ORR will be presented as the point estimate together with the exact 95% CI according to the Clopper-Pearson method. The duration of response (DoR) and progression-free survival (PFS) will be presented for all patients in Part 2, summarized using the Kaplan-Meier (K-M) method with associated K-M curves. The median DoR and PFS will be presented, as well as the rates at clinically relevant time points, together with the associated 95% CIs.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study-specific procedures
* Females and males >/= 18 years
* Primary diagnosis of NSCLC with evidence of disease progression during or following treatment with an EGFR tyrosine kinase inhibitor (diagnosis of NSCLC that is confirmed by cytology is acceptable)
* Willing to undergo tumor biopsy (e.g., excision, core biopsy, or endoscopic biopsy), preferably of a progressing lesion, and provide blood and urine for biomarker testing
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study
* Prior treatment with osimertinib or another T790M directed therapy
* Current participation in another clinical study with an investigational product or patients who plan to receive any treatment that is not FDA-approved for EGFR mutation positive NSCLC at any time during the course of this study
* Use of any chemotherapeutic agent within 1 week of tissue, plasma, and urine sample collection
* For women - currently pregnant or plan to become pregnant during the course of the study: pre-menopausal women of childbearing potential must have a urine or serum pregnancy test performed during the screening/enrollment period and prior to initiating anti-cancer treatment
* Judgment by the investigator that the patient should not participate in the study due to the patient being unlikely to comply with study procedures, restrictions, and requirements, such as in the case of severe or uncontrolled systemic disease.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for this trial is non-small cell lung cancer patients who will come primarily from the community oncology practice setting.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2018-11-10 (Actual)

PRIMARY OUTCOMES:
The percentage of patients whose T790M results on Trovera urine AND Guardant360 plasma testing match their T790M results on cobas tissue testing. | Visit 1 (Day-21 to Day 0)
  The Overall Percent Agreement will be estimated as analytic concordance between Guardant360 plasma and Trovera urine testing versus cobas tissue testing in identifying T790M status (positive or negative). The Positive Percent Agreement will be estimated as the percentage of cobas tissue positive patients who are also Guardant360 plasma and/or Trovera urine positive. The Negative Percent Agreement will be estimated as the percentage of cobas tissue negative patients who are also Guardant360 plasma and Trovera urine negative.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Every 12 weeks for 12 months
  The number of patients achieving a confirmed partial response or complete response per RECIST 1.1 from treatment with osimertinib.
Duration of Response (DoR) | Every 12 weeks for the first 12 months, then at week 72
  The time from first documented tumor response defined by RECIST 1.1 from osimertinib treatment until the date of documented progression or death from any cause.
Progression Free Survival (PFS) | Every 12 weeks for the first 12 months, then at Week 72
  Defined as the time from date of first dose of osimertinib until the date of disease progression by RECIST 1.1 or death by any cause.

OTHER OUTCOMES:
Number of procedure-related adverse events and Serious Adverse Events (SAEs) | Up to 8 weeks after Visit 1
  To evaluate safety and tolerability of study procedures.
Percentage of patients whose Trovera urine OR Guardant360 plasma T790M results are the same as their cobas tissue T790M results. | Visit 1 (Day -21 to Day 0)
  The overall percent agreement will be estimate as analytic concordance between cobas tissue and Guardant360 plasma, and cobas tissue and Trovera urine testing in identifying T790M status. The positive percent agreement will be estimated as the percentage of cobas tissue positive patients who are also Guardant360 plasma positive and cobas tissue positive patients who are Trovera urine positive. The negative percent agreement will be estimated as the percentage of cobas tissue negative patients who are also Guardant360 plasma negative and cobas tissue negative patients who are Trovera urine negative.
The presence of additional biomarkers from the blood and/or urine of NSCLC patients who have progressed during or following treatment with an EGFR tyrosine kinase inhibitor | Visit 1 (Day -21 to Day 0)
  Biomarker results will be assessed and may be compared to T790M status and/or clinical response.
Percentage of patients whose Trovera urine OR Guardant360 plasma EGFR mutation results are the same as their cobas tissue EGFR mutation results. | Visit 1 (Day -21 to Day 0)
  The overall percent agreement will be estimated as analytic concordance between Guardany360 plasma and Trovera urine testing versus cobas tissue testing in identifying the status of specified EGFR mutations. The positive percent agreement will be estimated as the percentage of cobas tissue positive patients who are also Guardant360 plasma and/or Trovera urine positive. The negative percent agreement will be estimated as the percentage of cobas tissue negative patients who are also Guardant360 plasma and Trovera urine negative.
Physical Exam | Up to 8 weeks after Visit 1
  Changes in physical exams from baseline
Vital signs | Up to 8 weeks after Visit 1
  Changes in vital signs from baseline
ECG | Up to 8 weeks after Visit 1
  Changes in ECGs from baseline.
Number of Adverse Events, Serious Adverse Events, and Adverse Events of Special Interest | From the time of first dose of osimertinib through 30 days past the last dose of osimertinib or 30 days after Week 72, if osimertinib treatment remains ongoing at Week 72.
  To evaluate the safety and tolerability of osimertinib.
Physical Exam | From the time of first dose of osimertinib through the date of last dose of osimertinib or at Week 72, whichever comes first.
  To evaluate the safety and tolerability of osimertinib.
Vital signs | From the time of first dose of osimertinib through the date of last dose of osimertinib or at Week 72, whichever comes first.
  To evaluate the safety and tolerability of osimertinib
ECG | From the time of first dose of osimertinib through the date of last dose of osimertinib or at Week 72, whichever comes first.
  To evaluate the safety and tolerability of osimertinib

CONTACTS AND LOCATIONS:
Overall Officials: Nabil Chehab, PhD, Study Director — AstraZeneca
Locations (22):
- United States (19):
  - Research Site, Anaheim, California
  - Research Site, Los Angeles, California
  - Research Site, Santa Rosa, California
  - Research Site, St. Helena, California
  - Research Site, Deerfield Beach, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, Boise, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Harvey, Illinois
  - Research Site, Annapolis, Maryland
  - Research Site, Southfield, Michigan
  - Research Site, Brick, New Jersey
  - Research Site, Farmington, New Mexico
  - Research Site, White Plains, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Hendersonville, North Carolina
  - Research Site, Kettering, Ohio
  - Research Site, Seattle, Washington
- Canada (3):
  - Research Site, Edmonton, Alberta
  - Research Site, Newmarket, Ontario
  - Research Site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Molina JR, Yang P, Cassivi SD, Schild SE, Adjei AA. Non-small cell lung cancer: epidemiology, risk factors, treatment, and survivorship. Mayo Clin Proc. 2008 May;83(5):584-94. doi: 10.4065/83.5.584. PMID 18452692
- [Background] Morgillo F, Della Corte CM, Fasano M, Ciardiello F. Mechanisms of resistance to EGFR-targeted drugs: lung cancer. ESMO Open. 2016 May 11;1(3):e000060. doi: 10.1136/esmoopen-2016-000060. eCollection 2016. PMID 27843613
- [Background] Sullivan I, Planchard D. Osimertinib in the treatment of patients with epidermal growth factor receptor T790M mutation-positive metastatic non-small cell lung cancer: clinical trial evidence and experience. Ther Adv Respir Dis. 2016 Dec;10(6):549-565. doi: 10.1177/1753465816670498. Epub 2016 Oct 26. PMID 27784815
- [Background] Oxnard GR, Thress KS, Alden RS, Lawrance R, Paweletz CP, Cantarini M, Yang JC, Barrett JC, Janne PA. Association Between Plasma Genotyping and Outcomes of Treatment With Osimertinib (AZD9291) in Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2016 Oct 1;34(28):3375-82. doi: 10.1200/JCO.2016.66.7162. Epub 2016 Jun 27. PMID 27354477
- [Background] Thress KS, Brant R, Carr TH, Dearden S, Jenkins S, Brown H, Hammett T, Cantarini M, Barrett JC. EGFR mutation detection in ctDNA from NSCLC patient plasma: A cross-platform comparison of leading technologies to support the clinical development of AZD9291. Lung Cancer. 2015 Dec;90(3):509-15. doi: 10.1016/j.lungcan.2015.10.004. Epub 2015 Oct 9. PMID 26494259
- [Background] Kawamura T, Kenmotsu H, Taira T, Omori S, Nakashima K, Wakuda K, Ono A, Naito T, Murakami H, Mori K, Nakajima T, Ohde Y, Endo M, Takahashi T. Rebiopsy for patients with non-small-cell lung cancer after epidermal growth factor receptor-tyrosine kinase inhibitor failure. Cancer Sci. 2016 Jul;107(7):1001-5. doi: 10.1111/cas.12963. Epub 2016 Jun 21. PMID 27145431
- [Background] Lorenz J, Blum M. Complications of percutaneous chest biopsy. Semin Intervent Radiol. 2006 Jun;23(2):188-93. doi: 10.1055/s-2006-941449. PMID 21326762
- [Background] Reckamp KL, Melnikova VO, Karlovich C, Sequist LV, Camidge DR, Wakelee H, Perol M, Oxnard GR, Kosco K, Croucher P, Samuelsz E, Vibat CR, Guerrero S, Geis J, Berz D, Mann E, Matheny S, Rolfe L, Raponi M, Erlander MG, Gadgeel S. A Highly Sensitive and Quantitative Test Platform for Detection of NSCLC EGFR Mutations in Urine and Plasma. J Thorac Oncol. 2016 Oct;11(10):1690-700. doi: 10.1016/j.jtho.2016.05.035. Epub 2016 Jul 25. PMID 27468937
- [Background] Shyamala K, Girish HC, Murgod S. Risk of tumor cell seeding through biopsy and aspiration cytology. J Int Soc Prev Community Dent. 2014 Jan;4(1):5-11. doi: 10.4103/2231-0762.129446. PMID 24818087
- [Background] Goss G, Tsai CM, Shepherd FA, Bazhenova L, Lee JS, Chang GC, Crino L, Satouchi M, Chu Q, Hida T, Han JY, Juan O, Dunphy F, Nishio M, Kang JH, Majem M, Mann H, Cantarini M, Ghiorghiu S, Mitsudomi T. Osimertinib for pretreated EGFR Thr790Met-positive advanced non-small-cell lung cancer (AURA2): a multicentre, open-label, single-arm, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1643-1652. doi: 10.1016/S1470-2045(16)30508-3. Epub 2016 Oct 14. PMID 27751847
- [Background] Soria JC, Wu YL, Nakagawa K, Kim SW, Yang JJ, Ahn MJ, Wang J, Yang JC, Lu Y, Atagi S, Ponce S, Lee DH, Liu Y, Yoh K, Zhou JY, Shi X, Webster A, Jiang H, Mok TS. Gefitinib plus chemotherapy versus placebo plus chemotherapy in EGFR-mutation-positive non-small-cell lung cancer after progression on first-line gefitinib (IMPRESS): a phase 3 randomised trial. Lancet Oncol. 2015 Aug;16(8):990-8. doi: 10.1016/S1470-2045(15)00121-7. Epub 2015 Jul 6. PMID 26159065
- See also: Ferlay J, Soerjomataram I, Ervik M, et al. GLOBOCAN 2012 v1.0, Cancer Incidence and Mortality Worldwide: IARC CancerBase No. 11 [Internet]. Lyon, France: International Agency for Research on Cancer; 2013. Accessed on 18 January 2017. — http://globocan.iarc.fr
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160L00032&attachmentIdentifier=cd46d2b7-9a88-4ec4-a9db-0d67b90ad64a&fileName=D5160L00032_CSR_v1.0_synopsis-redacted.pdf&versionIdentifier=
- See also: redacted synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160L00032&attachmentIdentifier=cc8b5a53-37d2-420e-8d2d-ca6c09cfd801&fileName=D5160L00032_CSR_v1.0_synopsis-redacted.pdf&versionIdentifier=